CLINICAL TRIAL: NCT03252509
Title: Outpatient Percutaneous Radiologic Gastrostomy in Patients With Head and Neck Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: INCA RI
Record Dates: First submitted 2017-08-15; First posted 2017-08-17 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2018-03

CONDITIONS: Gastrostomy; Head and Neck Neoplasms; Malignant Neoplasm
Keywords: percutaneous radiologic gastrostomy; Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: Pre a post interventional study, in patients with head and neck neoplasms, eligible for an outpatient procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Percutaneous radiologic gastrostomy. (Experimental): Outpatient percutaneous radiologic gastrostomy in patients with head and neck tumors before, during or after the oncologic treatment.
  Interventions: Procedure: Percutaneous radiologic gastrostomy

INTERVENTIONS:
Procedure: Percutaneous radiologic gastrostomy — Percutaneous radiologic gastrostomy: Under conscious sedation and local analgesia, the ultrasound is performed to determine abdominal structures. The stomach is distended using room air through a nasogastric catheter or a 5 French (Fr) catheter. Gastropexy is performed under fluoroscopic guidance. The stomach is accessed using a 18 gauge (G) needle. Guidewire is advanced to the stomach. Progressive tract dilatations until the size of the gastrostomy tube is achieved. The catheter is advanced through the peel-away sheath. The catheter's balloon is inflated with 10ml of distilled water. Iodine contrast is injected to confirm position. After the procedure, the patient is observed for 3 hours. If there are no complications, the patient is discharged.

SUMMARY:
This study intends to evaluate the security and success rate of large bore percutaneous radiologic gastrostomy in patients with head and neck tumors, as a outpatient procedure.

DETAILED DESCRIPTION:
Percutaneous gastrostomy is a procedure that intends to provide prolonged alimentary access to patients with normal gastrointestinal tract, which are unable to eat or are facing troubles with deglutition.

Nowadays it is considered as the first line procedure to prolonged enteral access on this patients.

The indications to perform a percutaneous gastrostomy in a cancer center are usually related to head and neck, central nervous system and esophagus tumors. In our institution around 80% of the percutaneous gastrostomy are performed in patients with head an neck tumors.

Although percutaneous gastrostomy is considered a safe procedure, there are some complications related, specially in oncologic patients. Those complications are reported in about 40% of the cases.

Percutaneous gastrostomy is usually performed as a inpatient procedure, which leads to hospitalization costs. However, some studies have shown that is safe and viable to perform percutaneous gastrostomy (both endoscopic or radiologic), as a outpatient procedure, in patients with head a neck tumors.

As both techniques (endoscopic and radiologic) present similar results, patients treated in our institution that require a percutaneous gastrostomy are referred to endoscopic and interventional radiology departments.

Some of these patients are selected to undergo an outpatient procedure, based on social and clinical criteria.

The majority of the available data shows that both the endoscopic and the radiologic techniques present similar results in terms of security and rate of precocious and late complications, and that both are superior than the surgical technique, considering they are least invasive and related with lower rates of complication and costs.

In the present, the traction (Gauderer-Ponsky) technique is the most widely used in our institution for the endoscopic procedure.

In the interventional radiology department the percutaneous gastrostomy is performed using the introduction (Russel) technique, in which a guidewire is positioned after the stomach needle puncture, made under ultrasound or fluoroscopic guidance. After that, the tract is progressively dilated to allow the introduction of the gastrostomy balloon catheter, through the abdominal wall, using a peel-away sheath.

This same technique can be performed for the endoscopic gastrostomy, using the same gastrostomy kit, but under endoscopic guidance.

Some authors suggest that the introduction technique, although more challenging, is associated with less stoma infections, because is the only one that is not associated with oral catheterization.

For the patients with head an neck tumors, there is also a reduced risk of metastases implants on the puncture site.

Besides those considerations, the data available is still not consensual.

ELIGIBILITY:
Inclusion Criteria:

* Surgical risk ASA I-III, Karnofsky Performance Status >70, acceptance and comprehension of the orientations and after-care, adequate social a familiar support, easy access to the hospital.

Exclusion Criteria:

* patients who live more than one hour away from the hospital, coagulopathies, refuse to join the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Complication rate. | Up to 24 weeks.
  Rate of other complications like bleeding, infection, cutaneous fistulae.

SECONDARY OUTCOMES:
Duration of gastrostomy. | Up to 24 weeks.
  Duration of primary gastrostomy tube.
Technical success rate. | Immediately.
  Gastrostomy tube insertion into gastric lumen.
Procedure duration time. | Immediately after the procedure.
  Time necessary to place the gastrostomy tube, from gastric distention to local dressing.
Pain intensity. | Immediately after the procedure and during the total follow-up period - Up to 24 weeks.
  Pain will be measured according to pain score (1-10).
Additional procedures. | Up to 24 weeks.
  Procedures required after gastrostomy placement, like tube reinsertion or tube changes.

OTHER OUTCOMES:
Gastrostomy outcomes after the follow-up period. | Up to 24 weeks.
  Death for any reason using the gastrostomy tube, elective withdrawal after recovery of swallow function and persistence with gastrostomy tube.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo R Gouveia, Principal Investigator — Instituto Nacional do Câncer
Locations (1):
- Instituto Nacional do Cancer - HC1, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Campoli PM, Cardoso DM, Turchi MD, Ejima FH, Mota OM. Assessment of safety and feasibility of a new technical variant of gastropexy for percutaneous endoscopic gastrostomy: an experience with 435 cases. BMC Gastroenterol. 2009 Jun 26;9:48. doi: 10.1186/1471-230X-9-48. PMID 19558672
- [Background] Cantwell CP, Perumpillichira JJ, Maher MM, Hahn PF, Arellano R, Gervais DA, Mueller PR. Antibiotic prophylaxis for percutaneous radiologic gastrostomy and gastrojejunostomy insertion in outpatients with head and neck cancer. J Vasc Interv Radiol. 2008 Apr;19(4):571-5. doi: 10.1016/j.jvir.2007.11.012. PMID 18375303
- [Background] Cosentini EP, Sautner T, Gnant M, Winkelbauer F, Teleky B, Jakesz R. Outcomes of surgical, percutaneous endoscopic, and percutaneous radiologic gastrostomies. Arch Surg. 1998 Oct;133(10):1076-83. doi: 10.1001/archsurg.133.10.1076. PMID 9790204
- [Background] Foster JM, Filocamo P, Nava H, Schiff M, Hicks W, Rigual N, Smith J, Loree T, Gibbs JF. The introducer technique is the optimal method for placing percutaneous endoscopic gastrostomy tubes in head and neck cancer patients. Surg Endosc. 2007 Jun;21(6):897-901. doi: 10.1007/s00464-006-9068-9. Epub 2006 Dec 16. PMID 17180272
- [Background] Gauderer MW, Ponsky JL, Izant RJ Jr. Gastrostomy without laparotomy: a percutaneous endoscopic technique. J Pediatr Surg. 1980 Dec;15(6):872-5. doi: 10.1016/s0022-3468(80)80296-x. PMID 6780678
- [Background] Giordano-Nappi JH, Ishioka S, Maluf-Filho F, Hondo FY, Matuguma SE, Sakai P. A new device for the introducer technique for percutaneous endoscopic gastrostomy placement. Endoscopy. 2007 Feb;39 Suppl 1:E274-5. doi: 10.1055/s-2007-966615. Epub 2007 Oct 24. No abstract available. PMID 17957639
- [Background] Hiki N, Maetani I, Suzuki Y, Washizawa N, Fukuda T, Yamaguchi T; Tokyo Standard PEG Study Group. Reduced risk of peristomal infection of direct percutaneous endoscopic gastrostomy in cancer patients: comparison with the pull percutaneous endoscopic gastrostomy procedure. J Am Coll Surg. 2008 Nov;207(5):737-44. doi: 10.1016/j.jamcollsurg.2008.06.335. Epub 2008 Aug 9. PMID 18954787
- [Background] Horiuchi A, Nakayama Y, Tanaka N, Fujii H, Kajiyama M. Prospective randomized trial comparing the direct method using a 24 Fr bumper-button-type device with the pull method for percutaneous endoscopic gastrostomy. Endoscopy. 2008 Sep;40(9):722-6. doi: 10.1055/s-2008-1077490. Epub 2008 Sep 4. PMID 18773341
- [Background] Koide T, Inamori M, Kusakabe A, Uchiyama T, Watanabe S, Iida H, Endo H, Hosono K, Sakamoto Y, Fujita K, Takahashi H, Yoneda M, Tokoro C, Yasuzaki H, Goto A, Abe Y, Kobayashi N, Kubota K, Saito S, Nahajima A. Early complications following percutaneous endoscopic gastrostomy: results of use of a new direct technique. Hepatogastroenterology. 2010 Nov-Dec;57(104):1639-44. PMID 21443135
- [Background] Kusaka K, Itoh T, Kawaura K, Yamakawa J, Takahashi T, Kanda T. Three-point fixation of stomach to abdominal wall in the percutaneous endoscopic gastrostomy procedure. Endoscopy. 2005 May;37(5):494. doi: 10.1055/s-2005-861233. No abstract available. PMID 15844032
- [Background] Maetani I, Tada T, Ukita T, Inoue H, Sakai Y, Yoshikawa M. PEG with introducer or pull method: a prospective randomized comparison. Gastrointest Endosc. 2003 Jun;57(7):837-41. doi: 10.1016/s0016-5107(03)70017-0. PMID 12776029
- [Background] de Souza e Mello GF, Lukashok HP, Meine GC, Small IA, de Carvalho RL, Guimaraes DP, Mansur GR. Outpatient percutaneous endoscopic gastrostomy in selected head and neck cancer patients. Surg Endosc. 2009 Jul;23(7):1487-93. doi: 10.1007/s00464-009-0381-y. Epub 2009 Mar 5. PMID 19263126
- [Background] Russell TR, Brotman M, Norris F. Percutaneous gastrostomy. A new simplified and cost-effective technique. Am J Surg. 1984 Jul;148(1):132-7. doi: 10.1016/0002-9610(84)90300-3. PMID 6430111
- [Background] Rustom IK, Jebreel A, Tayyab M, England RJ, Stafford ND. Percutaneous endoscopic, radiological and surgical gastrostomy tubes: a comparison study in head and neck cancer patients. J Laryngol Otol. 2006 Jun;120(6):463-6. doi: 10.1017/S0022215106000661. PMID 16772054
- [Background] Sacks BA, Vine HS, Palestrant AM, Ellison HP, Shropshire D, Lowe R. A nonoperative technique for establishment of a gastrostomy in the dog. Invest Radiol. 1983 Sep-Oct;18(5):485-7. doi: 10.1097/00004424-198309000-00015. PMID 6642944
- [Background] Tucker AT, Gourin CG, Ghegan MD, Porubsky ES, Martindale RG, Terris DJ. 'Push' versus 'pull' percutaneous endoscopic gastrostomy tube placement in patients with advanced head and neck cancer. Laryngoscope. 2003 Nov;113(11):1898-902. doi: 10.1097/00005537-200311000-00007. PMID 14603043
- [Background] Van Dyck E, Macken EJ, Roth B, Pelckmans PA, Moreels TG. Safety of pull-type and introducer percutaneous endoscopic gastrostomy tubes in oncology patients: a retrospective analysis. BMC Gastroenterol. 2011 Mar 16;11:23. doi: 10.1186/1471-230X-11-23. PMID 21410958
- [Background] Walton GM. Complications of percutaneous gastrostomy in patients with head and neck cancer--an analysis of 42 consecutive patients. Ann R Coll Surg Engl. 1999 Jul;81(4):272-6. PMID 10615198
- [Background] Wilhelm SM, Ortega KA, Stellato TA. Guidelines for identification and management of outpatient percutaneous endoscopic gastrostomy tube placement. Am J Surg. 2010 Mar;199(3):396-9; discussion 399-400. doi: 10.1016/j.amjsurg.2009.08.023. PMID 20226918
- [Background] Wollman B, D'Agostino HB. Percutaneous radiologic and endoscopic gastrostomy: a 3-year institutional analysis of procedure performance. AJR Am J Roentgenol. 1997 Dec;169(6):1551-3. doi: 10.2214/ajr.169.6.9393163.